CLINICAL TRIAL: NCT01181739
Title: The Effect of Experience and Training on the Accuracy of CT (Computed Tomography) Colonography in Comparison With Optical Colonoscopy in the Detection of Colonic Neoplasia
Brief Title: Computed Tomography (CT) Colonography Versus Optical Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Society of Intestinal Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: H08-00776
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Colonic Neoplasia
Keywords: Colonoscopy; Virtual Colonoscopy; Colonography; Colorectal Cancer; Colonic Polyps; Screening
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Colonic Mucosal Biopsy specimens obtained at the time of colonoscopy
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to compare traditional Colonoscopy with CT Colonography, commonly known as "virtual colonoscopy". The study will compare the ability of both procedures as screening tests to identify polyps in the colon in patients at average risk for developing polyps. The patient preferences for each procedure will be assessed by means of a standardized questionnaire. As well the ability observers with differing levels of experience to read the CT scans and detect polyps will be compared. All patients will receive both CT scans and traditional colonoscopy on the same day.

DETAILED DESCRIPTION:
1. Purpose To study the Effect of Experience and Training on the Accuracy of CT (Computed Tomography) Colonography in Comparison with Optical Colonoscopy in the Detection of Colonic Neoplasia

2. Hypotheses

1. The accuracy (sensitivity and specificity) of interpretation of the CTC images will improve with each 100 scans examined. Less time will be required to interpret the CTC images after each successive 100 scans. The accuracy of each of the observers will be similar.
2. The sensitivity and specificity will be similar for CTC and OC for the last 100 patients undergoing both examinations.
3. Patients will prefer CTC to OC based on comfort and ease of the procedure.
4. CTC will have the added benefit of identifying extra-colonic findings which will not be found on OC. CTC will be performed at a lower cost per patient with a lower complication rate than for OC and will take a similar amount of time to perform.

3. Justification Screening is believed to decrease the incidences of colorectal cancer and death as a result of the detection of both precancerous lesions and cancers at early stages4-6. Fecal occult blood testing and flexible sigmoidoscopy can miss a substantial number of significant lesions7. Despite its risk, inconvenience, and cost, optical colonoscopy is the primary screening tool for colorectal cancer when performed every 10 years, beginning at 50 years of age in people who are at average risk8,9. Screening is also recommended at a younger age for populations at increased risk10.

Virtual colonoscopy is a rapidly evolving technique in which data from computed tomography (CT) is used to generate both two-dimensional and three-dimensional displays of the colon and rectum. This minimally invasive method for the examination of the colon, also referred to as CT colonography (CTC), is a promising alternative to optical colonoscopy for use in widespread screening, as it requires no intravenous administration of sedatives or analgesia and little recovery time.

Many studies have sought to compare the utility of CTC and optical colonoscopy (OC) in the detection of colonic polyps and adenocarcinomas in various patient populations.

Before CTC can be used in usual practice the training required by those interpreting the studies needs to be further studied so that guidelines can be created defining requirements necessary prior to implementation of this screening strategy.

4. Study Objectives: To determine the effects of previous training and experience on the accuracy of polyp and cancer detection for CTC in patients at above average risk for colorectal cancer.

1. To assess the learning curve of GI radiologists (experienced and not experienced with CTC interpretation), a GI fellow and a family physician as they acquire experience in reading CTC datasets by measuring the detection rates, miss rates and the amount of time needed to read images for the 1st, 2nd and 3rd set of 100 CTC's which they interpret.
2. The study will also determine the sensitivity and specificity of CTC compared with OC for the detection of colonic polyps (of various sizes) and adenocarcinoma in patients at high risk for colorectal cancer (those over 45 years of age with a family history of colorectal cancer, those with positive screening tests and those with suggestive symptoms).
3. Patient satisfaction with both CTC and OC will be evaluated by means of a patient questionnaire.
4. The two procedures will be compared in terms of complication rates, the time required to perform each test, extra-colonic findings and the cost to perform each procedure per patient.

5. Research Method A non-randomized, evaluator blinded study of 300 consecutive patients at high risk for colonic neoplasia referred for colonoscopy. Each patient is to undergo standard colonoscopy preparation on the day prior to CT Colonography (CTC) followed within 2 hours by optical colonoscopy (OC). Patients will be men and women aged 19 - 65 years who were scheduled to undergo elective colonoscopy referred from a suburban primary care setting.

Study population The study participants will consist of two main populations. The first will include patients at average to high risk of colonic neoplasia who are eligible for screening colonoscopy. Average risk patients are those aged 45-65 who wish to undergo screening for colorectal cancer. High risk patients include those with a family history of colorectal cancer, previous colorectal cancer or neoplasia, positive screening tests (Fecal Occult Blood (FOBT), flexible sigmoidoscopy, digital rectal exam or air contrast barium enema) and patients with gastrointestinal symptoms and signs (abdominal pain, rectal bleeding, anemia). Patients will be recruited from a suburban primary care medical clinic in Coquitlam, B.C. (North Road Medical Centre) and referred to a gastroenterology clinic in downtown Vancouver (Pacific Gastroenterology Associates) or recruited from the gastroenterology clinic directly.

Ethical approval will be obtained from the University of British Columbia and the St. Paul's Hospital Institutional Review Boards. A study investigator will obtain informed consent from potential study participants.

Design After obtaining informed consent, participants will be instructed to consume a clear liquid diet for the 24 hours prior to the exam. Patients will receive detailed instructions regarding bowel preparation using oral Picosalax and Bisacodyl suppositories to be taken on the day prior to their procedures (see Appendix 2). Instructions will also be provided regarding the intake of oral barium and gastrograffin which will be used as stool tagging agents (see Appendix 2). As both CTC and OC will take place on the same day, the preparation will be identical for both procedures. No sedative agents will be administered during CTC. Colonic distention for CTC will be achieved with automated low-pressure delivery of carbon dioxide. Patients will be allowed sips of clear fluid on the morning of the examinations and will then be kept without oral intake until after both CTC and OC are completed.

CT Colonography Patients will be given an appointment time for presentation to St. Paul's Hospital radiology department. After reporting, they will be asked to change into a hospital gown and CT scanning will be performed. Images will be acquired using the GE Lightspeed 64 row multidetector CT scanner. Slices will be obtained at 0.75mm resolution and will be reconstructed using GE Healthcare software at a resolution of 1.25mm. Scans will be obtained during a single breath hold using a low radiation exposure protocol (~30-50 mAs which corresponds to an absorbed radiation dose of 3-5 mSv). The quality and adequacy of the images will be assessed before patients leave the radiology department to await colonoscopy which will be performed within 2 hours.

Interpretation There will be 2 radiologist readers both experienced in gastrointestinal imaging and one of whom is experienced in CTC interpretation. The Radiologists will review the scans and record their findings in 4 separate envelopes, one for each section of the colon (rectum and sigmoid, descending, transverse and right colon). The size of lesions found will be recorded from the optimum view using electronic callipers. Finally, the radiologists will review the films for any extra-colonic findings that will be recorded separately. Similarly, a GI Fellow and a Family Physician will review the scans recording their findings in the same manner. However, at least one Radiologist will review the films at the time of the examination to ensure that they are of adequate quality and to provide their interpretation prior to OC. The amount of time taken to read the films for each reviewer will be recorded as a total time to read all views for each patient. Observers will be made aware of optical colonoscopy results after each 100 procedures.

Optical Colonoscopy Within 2 hours of finishing the CTC imaging, participants will undergo OC with conscious sedation using a combination of midazolam and Demerol or fentanyl to achieve patient comfort. An experienced gastroenterologist using an Olympus colonoscope will perform the colonoscopies. The endoscopist, blinded to the CTC results will examine the colon on withdrawal of the endoscope, recording findings for each of the four segments of the colon. Each segment is then to be sequentially unblinded allowing the endoscopist to review the Radiologists findings for each colonic segment on CTC. Polyps detected at endoscopy will be removed using standard techniques (biopsy forceps or snare cautery) and submitted for pathological assessment.

Advanced neoplasms will be divided by pathology into adenocarcinomas and polyps. Polyps will be further categorized according to size (≤5mm, 6-9mm and ≥10mm). Morphologic characteristics of the lesions will also be recorded by viewers as sessile, pedunculated or flat. Lesion size is to be determined by measurement of removed lesions (before fixation) or estimated at endoscopy by comparison to the biopsy forceps, for those lesions that are not removed.

Patient Questionnaires Following endoscopy, patients will be transferred to recovery area where they will undergo monitoring of their vital signs following standard practice guidelines, until they are ready for discharge. Immediately prior to discharge, patients will be given a 10 question written survey, for self-completion (see appendix 1). The recovery room nurse will give this to them after final consultation with the Gastroenterologist while in the recovery room. Patients will be given as much time as necessary to complete the survey and instruction to seal the survey in an envelope and return it to the nurse prior to leaving the recovery room.

In order to assess the test/retest reliability of the survey, a random sample of patients will be mailed a second survey (identical to the first) 3 - 4 weeks after the day of examination. Enclosed will be instructions for self-completion of the survey and a self addressed, postage paid, return envelope to allow for its return.

6. Statistical Analysis The reference standard of polyp detection will be the results of OC after each colonic segment is re-examined once the CTC results are known. Tests of accuracy will be sensitivity, specificity, true positive and true negative results with comparison to the reference standard. ROC curves for CTC and OC will be derived after all tests are completed. The AUC for each tests' ROC curve will be used to compare accuracy between these two tests. ROC curves and the AUC statistic will be derived from the dataset once divided according to each 100 CTC performed and by each reader to evaluate the learning curve of this test. Tests of significance will be McNemar's test, paired t-tests, and chi-square tests as appropriate. Interobserver reliability will be reported as a kappa statistic.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 65 years of age
* Have a recognized indication for optical colonoscopy, including high risk for colorectal cancer
* Over 45 years of age with a family history of colorectal cancer, those with positive screening tests (FOBT, DRE, flexible sigmoidoscopy and contrast enema)
* Previous history of advanced adenomas and those with suggestive symptoms and signs (bleeding, abdominal pain, anemia)
* Must be able to read and understand English and must be able to give informed consent

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 19 - 65 years of age at with a recognized indication for optical colonoscopy, including those high risk for colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
CT colonography | During procedure
  CT colonography (CTC), is a promising alternative to optical colonoscopy for use in widespread screening, as it requires no intravenous administration of sedatives or analgesia and little recovery time.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enns, Dr., Principal Investigator — University of British Columbia; Jacquie Brown, Dr., Study Director — University of British Columbia; Jennifer Telford, Dr., Study Director — University of British Columbia; Gregory Rosenfeld, Dr., Study Director — University of British Columbia; Pari Tiwari, Dr., Study Director — University of British Columbia; Darin Krygier, Dr., Study Director — University of British Columbia; Brian Bressler, Dr., Study Director — University of British Columbia; Patrick Vos, Dr., Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Pacific Research Institute, Vancouver, British Columbia